CLINICAL TRIAL: NCT05037812
Title: Determining the Role of Periarticular Multimodal Analgesia in Decreasing Perioperative Pain in Tibial Plateau Fractures
Brief Title: Role of Multimodal Analgesia in Decreasing Perioperative Pain in Tibial Plateau Fractures
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Justin Haller, Principle Investigator, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117178
Record Dates: First submitted 2021-09-02; First posted 2021-09-08 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Tibial Plateau Fractures
Keywords: Tibial Plateau Fractures; Periarticular Multimodal Analgesia; Perioperative Pain
MeSH Terms: conditions — Tibial Plateau Fractures | interventions — Sodium Chloride; Morphine; Epinephrine; Clonidine; Ketorolac Tromethamine; Ketorolac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Saline injection (Placebo Comparator): Saline
  Interventions: Drug: Saline injection
- Multimodal injections (Experimental): Superficial multimodal analgesia composition includes 5mg morphine, 500 micrograms epinephrine, and 4ml normal saline.
  Deep medial multimodal analgesia composition includes 2.5mg morphine, 40 micrograms clonidine, 15mg ketorolac, and 4ml normal saline.
  Interventions: Drug: Multimodal injections

INTERVENTIONS:
Drug: Saline injection — Saline
  Other Names: 0.9%NaCl (sodium chloride) H2O (saline)
  Arms: Saline injection
Drug: Multimodal injections — 5mg morphine, 500 micrograms epinephrine, and 4ml normal saline (superficial injection).
  2.5mg morphine, 40 micrograms clonidine, 15mg ketorolac, and 4ml normal saline (deep injection).
  Other Names: Morphine sulfate (MS) Contin, Astramorph, Depodur, Duramorph, Infumorph, Kadian, MorphaBond, Arymo ER (morphine); Adrenalin (epinephrine); Catapres, Kapvay (clonidine); Toradol (ketorolac); 0.9%NaCl (sodium chloride) H2O (saline)
  Arms: Multimodal injections

SUMMARY:
The investigators goal of the proposed research study is to determine the effectiveness of periarticular multimodal analgesia in the setting of tibial plateau fractures. Effectiveness of the multimodal analgesia is defined as lower pain scores.

DETAILED DESCRIPTION:
Pain control in the setting of orthopaedic trauma has always been imperative for patient comfort and to enhance functional recovery. However, the current opioid epidemic makes effective pain control even more critical. Furthermore, the Center of Medicare and Medicaid Services have developed tools for rating physician care, of which, pain control is considered a contributing part. The operative management of tibial plateau fractures requires adequate pain control to allow for early motion of the joint. Recently, multimodal pain therapy has been proposed as way to accomplish effective postoperative pain relief. This is difficult for this injury as any form of regional analgesia such as nerve blocks are not possible due to the possibility of compartment syndrome. The goal of the proposed research study is to determine the effectiveness of periarticular multimodal analgesia in the setting of tibial plateau fractures. Effectiveness of the multimodal analgesia is defined as lower pain scores and decreased narcotic intake in the perioperative setting.

The expected outcomes of the study are based on the extensive total knee arthroplasty literature that shows decreased pain and narcotic usage in the peri-operative period with peri-articular multimodal analgesia injections. Furthermore, a recent study by other investigators showed decreased pain and narcotic usage in the first post-operative day following femur fractures of any kind. These data display the promise for the use of peri-articular multimodal analgesia in the setting of tibial plateau fractures.

With the rise of patient-centered care and outcome driven reimbursement, pain control is one of the main factors in both these domains. The Center for Medicaid and Medicare Services has developed the Total Performance Score for Hospitals, which is factored into the reimbursement for provided services. Pain Management is one of the main contributors to the score. Moreover, pain control has been shown to improve patient satisfaction, which is of increasing importance in medicine today.

While some lower extremity fractures can be managed with a nerve block, tibial plateau fractures have a significant risk of developing compartment syndrome that preclude these patients from receiving a nerve block as it does not allow clinical monitoring. As such, the remaining options are to control pain with IV and oral narcotics.

There is no data on the effectiveness of peri-articular multimodal analgesia for tibial plateau fractures. The majority of evidence behind these injections in reducing peri-operative pain and decreasing narcotic use comes from the total knee arthroplasty literature. Numerous studies have investigated the effect of these injections and shown a decrease in perioperative pain and use of perioperative narcotics.

Investigators have looked at multimodal analgesia injections in femur fractures of all kinds. The investigators found that in patients receiving the injection, their pain was decreased over the first postoperative day along with consuming fewer narcotics over the same time frame. Unfortunately, the randomization in these studies resulted in an unequal distribution of injuries that may have biased the results. The investigators noted, "further investigations are required to establish the efficacy of this multimodal protocol for the individual surgical procedures considered". Five patients with tibial plateau fractures have experimentally been treated with a local multimodal analgesia at the applying institution. All five have had a subjectively decreased amount of pain with no evidence of peroneal nerve palsy, compartment syndrome, or infection. If the proposed study finds similar results in decreasing pain and narcotic use, not only would patients have an overall better experience, but this would also help in decreasing narcotic related adverse events in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients who present with isolated tibial plateau fractures treated by the investigators
* English or Spanish speaking

Exclusion Criteria:

* Poly trauma injuries
* Any allergies to the medication used in the injections
* Significant head trauma (loss of consciousness, Glasgow Coma Scale (GCS)<15, brain bleed) that interferes with the ability to provide informed consent.
* Non-English or Non-Spanish Speaking

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2019-03-25 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) pain | Pre-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 4-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 8-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 12-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 16-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 20-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)
Visual Analog Scale (VAS) pain | 24-hours post-operative
  VAS pain score (0 no pain - 10 severe pain)

CONTACTS AND LOCATIONS:
Overall Officials: Justin Haller, MD, Principal Investigator — University of Utah Orthopaedics
Locations (1):
- University of Utah Orthopaedic Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No